CLINICAL TRIAL: NCT07250100
Title: The Role of Microbiota in Pancreatic Cancer and Precursor Lesions
Acronym: MICROPAC
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Bojan Kovacevic, MD, ph.d., Herlev Hospital
Other Study IDs: H-22019595
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer; Microbiome
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pancreatic biopsies, oral swab, fekal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients suspected of pancreatic cancer
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Aprox. 300 patients suspected of pancreatic cancer. Of those, minimum of 50 patients with histologically confirmed PDAC in each of the stages I-II, III and IV, as some of the participants will be diagnosed with a non-malignant disease and will constitute the control group.

SUMMARY:
This is a prospective observational study aiming to investigate the microbiome in patients suspected of having pancreatic cancer. The purpose is to enhance diagnostic accuracy by developing screening protocols for high-risk individuals, identifying specific microbial biomarkers, and improving prognostic criteria to optimize treatment response.

Participants will be asked to complete a questionnaire, provide oral and fecal swabs, and-if clinically indicated-1-2 pancreatic biopsies will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a suspected lesion (solid/cystic) in the pancreas undergoing diagnostic or therapeutic endoscopic procedure
* Age of 18 years or above
* Signed informed consent form

Exclusion Criteria:

* Contraindications for endoscopic or surgical procedure, such as uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at Herlev Hospital or Rigshospitalet, who meets the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Composition of microbiota in pancreatic cancer | 2037
  To examine the composition of microbiota in pancreatic cancer and its precursors, to explore association between bacterial/fungal genera and final diagnosis, survival and risk of recurrence, but also to examine a possible role of microbiota in development of surgical adverse events.

SECONDARY OUTCOMES:
Databank | 2037
  To establish a databank containing clinical and demographic information from patients undergoing endoscopic evaluation of a pancreatic lesion
Biobank | 2037
  To establish a biobank of various biological material, herein tissue biopsies and/or cyst fluid, oral and fecal swabs at the time of inclusion and following end of therapy
Intratumor and gut mikrobiota | 2037
  To assess possible differences between intratumor and gut microbiota, and to inspect any changes in gut microbiota composition following surgery.
Intratumor viral DNA | 2037
  To investigate prevalence of intratumor viral DNA for the first time.
Microbiome-tumor interaction | 2037
  To elucidate microbiome-tumor interaction by examining intratumor gene expression and metabolism through RNA sequencing and isothermal microcalorimetry.
Microbiome composition | 2037
  To visualize microbiome composition within the tumor through fluorescence in situ hybridization confocal laser scanning microscopy and to determine geographic spread of the microbiome and its interaction with tumor cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev og Gentofte Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided